CLINICAL TRIAL: NCT01354015
Title: Diabetes Remote Care Management System
Acronym: DRMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University School of Medicine (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Vivian Fonseca, Professor, Tulane University School of Medicine
Organization: Tulane University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-Fonseca
Record Dates: First submitted 2011-05-06; First posted 2011-05-16 (Estimated); Results first posted 2015-01-13 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-03

CONDITIONS: Diabetes
Keywords: Diabetes; Technology
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Use of messaging system (Experimental): Use of DRMS
  Interventions: Device: DRMS
- Usual Care (No Intervention): Usual Care

INTERVENTIONS:
Device: DRMS — USE OF TEXT MESSAGING SYSTEM
  Arms: Use of messaging system

SUMMARY:
DRMS is a system that communicates with patients via text message using cellphones, computers and other devices. It reminds patients about multiple health care and disease related issues such as to test their blood sugars and send the result back to the system via text message. The system will then decided based on automated algorithms whether to send another message advising patients on changing their medication etc.

This pilot will enroll 100 injectible insulin dependent patients with uncomplicated Type 1 and Type 2 diabetes mellitus, using insulin, who will be enrolled to participate in the pilot. Patients will be randomized 1:1 to either DRMS or standard care. The patients in the DRMS program will undergo interactions with the system using multiple communications channels including cell phones, IVR, email, web and SMS messaging. The goals of the interactive programs are the following:

1. Monitor and intervene to remind patients to fill their prescriptions
2. Monitor and track insulin unit consumption utilization and timing of that dosage
3. Monitor and intervene when the patient does not use or take their medications as prescribed.
4. Monitor and track insulin unit consumption and timing of that dosage
5. Ask the patient for their glucose levels and then provide customized information to the patients regarding how to modify their medication to achieve the desired glucose level
6. Deliver automated dose adjustment directions based on the providers instructions
7. Coordinate personalized educational programs and messages into the automated intervention programs
8. Provide feedback to the patients, including performance and reinforcement to both providers and to patients.
9. Provide feedback to providers on patients performance as well as exception based reporting

The System will manage interventions in an automated fashion. Providers will intervene on an exception basis and only when automated interventions have not worked or the protocol requires immediate action by the provider. For example, if the glucose exceeds certain danger levels, as defined by the provider, a requirement might be to call and notify the doctor immediately.

DETAILED DESCRIPTION:
Primary Objective To determine the feasibility of using cell and phone technology to monitor, intervene and manage diabetes in patients using insulin.

Secondary Objectives:

1.To determine whether the DRMS system leads to improved glucose control (as measured by HgA1cHbA1c) during participation in the pilot

.2.To determine whether the DRMS system leads to improved management and adherence to insulin as well as other diabetic medications .3.To determine whether the DRMS system can be used as a cost effective solution for interventions across a broad segment (both demographic and economic groups) of the diabetes population.

This pilot will enroll 100 injectible insulin dependent patients with uncomplicated Type I1 and Type II2 diabetes mellitus, using insulin, who will be enrolled to participate in the pilot. Patients will be randomized 1:1 to either DRMS or standard care. It is anticipated that 150 patients will be screened in order to enroll 100 patients in the clinical trial. The patients in the DRMS program will undergo interactions with the system using multiple communications channels including cell phones, IVR, email, web and SMS messaging. The goals of the interactive programs are the following:

1. Monitor and intervene to remind patients to fill their prescriptions
2. Monitor and track insulin unit consumption utilization and timing of that dosage
3. Monitor and intervene when the patient does not use or take their medications as prescribed.
4. Monitor and track insulin unit consumption and timing of that dosage
5. Ask the patient for their glucose levels and then provide customized information to the patients regarding how to modify their medication to achieve the desired glucose level
6. Deliver automated titration directions based on the providers instructions
7. Coordinate personalized educational programs and messages into the automated intervention programs
8. Provide feedback to the patients, including performance and reinforcement to both providers and to patients.
9. Provide feedback to providers on patients performance as well as exception based reporting

The System will manage interventions in an automated fashion. Providers will intervene on an exception basis and only when automated interventions have not worked or the protocol requires immediate action by the provider. For example, if the glucose exceeds certain danger levels, as defined by the provider, a requirement might be to call and notify the doctor immediately.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older.
2. Able to read and understand the ICF and provide written consent.
3. Diagnosis of Type 1 or Type 2 diabetes. If Type 1 diabetes, requirement that they be on insulin and if Type 2 diabetes, requirement that they be on r insulin.
4. Recent HbA1c blood test (within the last 30 days).
5. An HbA1c reading of 7.5% - 9.0%.
6. Patient must own or have access to cell phone on a daily basis throughout the study period, and optionally can have a conventional phone or access to the Internet.
7. Patient possesses a blood sugar monitor and has access to supplies.
8. Patient is felt to be able to be compliant with the study.
9. Patient has no plans to move over the 6 month period of the study.

Exclusion Criteria:

1. Have active cancer other than basal cell carcinoma or cervical or breast cancer in situ.
2. In the opinion of the investigator are not suitable for entry into the study.
3. History of any psychiatric or neurologic condition that might impair the patient's ability to understand or to comply with the requirements of the study or to provide informed consent
4. Pregnant or breast-feeding females.
5. History (within last 6 months) of significant cardiovascular disease unless the disease is well-controlled. Significant cardiac diseases includes second/third degree heart block; clinically significant ischemic heart disease; QTcF interval > 450 msec at screening; poorly controlled hypertension; congestive heart failure of New York Heart Association (NYHA) Class II or worse (slight limitation of physical activity; comfortable at rest, but ordinary physical activity results in fatigue, palpitation, or dyspnea) or uncontrolled cardiac arrhythmias.
6. History of cerebrovascular accident (CVA) within 6 months prior to randomization or that resulted in ongoing neurologic instability.
7. Active infection or serious underlying medical condition (including any type of active seizure disorder within 12 months prior to randomization) that would impair the ability of the patient to participate in the trial.
8. Hypoglycemia Unawareness

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2011-05; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vivian Fonseca, Principal Investigator — Tulane University
Locations (1):
- Tulane University, New Orleans, Louisiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 01/01/12 from diabetes clinic
Period: Overall Study
Arm/Group | Use of Messaging System | Usual Care
Started | 50 | 48
Completed | 44 | 43
Not Completed | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Use of Messaging System | Usual Care | Total
Number analyzed (Participants) | 50 | 48 | 98
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.9 (10.3) | 59.3 (8.7) | 59.1 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 25 | 59
  Male | 16 | 23 | 39
Race/Ethnicity, Customized [Number; unit: participants] — self reported
  participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 1 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 37 | 27 | 64
    White | 13 | 17 | 30
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c
Description: change in A1c from baseline in intervention and control groups
Time Frame: baseline to 6 months
Population: Of the 50 enrolled in the Use of DRMS group, only 44 completed the visit at 6 months, and out of 48 enrolled in the Usual Care group only 43 completed the visit at 6 months. Therefore only those who completed the visit at 6 months were included in this analysis.
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Use of Messaging System | Usual Care
Number analyzed (Participants) | 44 | 43
Percent | -0.25 (0.2) | -0.4 (0.3)
Statistical Analysis 1: Comparison: Use of Messaging System; All statistical analysis used intent-to-treat methodology and all comparisons used a two-tailed test at the .05 level of significance. Continuous variables are reported as means and standard deviations. W; Test type: Superiority or Other; p = 0.2539, ANOVA; Mean Difference (Final Values) = 0.15, Standard Deviation 0.79

2. Secondary Outcome: Change in HbA1c Over 3 Months
Description: Change in HbA1c
Time Frame: baseline to 3 months
Population: Of the 50 enrolled in the Use of DRMS group, only 46 completed the visit at 3 months, and out of 48 enrolled in the Usual Care group only 45 completed the visit at 3 months. Therefore only those who completed the visit at 3 months were included in this analysis.
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Use of Messaging System | Usual Care
Number analyzed (Participants) | 46 | 45
Percent | -0.5 (0.3) | -0.2 (0.2)

ADVERSE EVENTS:
Arm/Group | Use of Messaging System | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/48
Other Adverse Events (participants affected / at risk) | 0/50 | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No